CLINICAL TRIAL: NCT02380300
Title: Registry Study of Clinical Application of MRI Compatible CIED
Status: Completed | Type: Observational
Sponsor: Biotronik (Beijing) Medical Device Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-01
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Need for MRI Imaging With Pacemaker or Implantable Cardioverter Defibrillator Implanted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to clear the Safety and Necessity of the Magnetic Resonance Imaging (MRI) in the Presence of CIEDs(Cardiovascular Implantable Electronic Devices).

ELIGIBILITY:
1. Inclusion criteria

   * Patient is >18 years old
   * Patient implanted with a Biotronik MRI compatible CIED (including the pacemaker, cardiac resynchronization therapy, implantable cardioverter defibrillator, and cardiac resynchronization therapy-defibrillator) in the past two months
   * Patient has provided a written informed consent
   * Patient's height is≥140cm
2. Exclusion criteria

   * Have other medical implants that may interact with MRI, e.g. abandoned pacemaker/ICD leads, lead extensions, mechanical valves, other active medical devices, non-MRI compatible devices
   * Life expectancy less than 2 years
   * Pregnant and/or breat-feeding females or females who intend to become pregnant in next two years
   * Patient is currently participating in another study
   * In the investigator's opinion patient will not be able to comply with the follow-up requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ProMRI CIED implanted，including ProMRI Pacemaker/CRT and ProMRI ICD/CRTD
Sampling Method: Non-Probability Sample
Enrollment: 2067 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Serious adverse events | two years
The raise of Impedance Threshold of the Atrial and Ventricle | immediate；one month
RA sensing amplitude (daily mean): < 1.5 mV or RV sensing amplitude (daily min.): < 2.0 mV | immediate；one month
The proportion of patients with CIED who need MRI examination | two years